CLINICAL TRIAL: NCT06008652
Title: A First-in-Human Multiple Expansion Cohort Phase 1 Study Evaluating the Safety and Activity of DR-0201 as Single Ascending Dose in Healthy Volunteers
Brief Title: A Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of DR-0201 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dren Bio (Industry)
Collaborators: Novotech (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DR-0201-HV-001
Record Dates: First submitted 2023-08-14; First posted 2023-08-23 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Healthy Adult Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DR-0201 (Experimental): Subjects in this arm will receive a single dose of DR-0201
  Interventions: Drug: DR-0201
- Placebo (Placebo Comparator): Subjects in this arm will receive a single dose of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DR-0201 — DR-0201 is a bi-specific antibody
  Arms: DR-0201
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled dose escalation study to evaluate the safety, tolerability, PK, PD, and immunogenicity of IV administered DR-0201 in healthy volunteers.

ELIGIBILITY:
Key Inclusion Criteria:

1. Healthy, in the opinion of the Investigator, as determined by medical evaluation including medical history, physical examination, laboratory tests, vital signs, and 12-lead ECGs. A subject with a clinical abnormality or laboratory parameter(s) outside the reference range for the population being studied that is not specifically listed in the inclusion or exclusion criteria may be included if the Investigator (in consultation with the Medical Monitor) agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures or data interpretation.
2. Between 18 and 55 years of age inclusive, at the time of signing the informed consent.
3. Body weight at screening ≥ 40 kg and < 120 kg, with body mass index between 18 and 30 kg/m2.
4. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form and in this protocol, including the protocol-mandate hospitalization.
5. Use of a highly effective contraceptive measure (< 1% failure rate; see Section 13.1) for all males and all females of childbearing potential during study and 90 days post dose for males and 30 days post dose for females. Females of childbearing potential need to have a confirmatory urine pregnancy test on Day -1. Females who are not of childbearing potential (i.e., who are considered to be post-menopausal [≥ 12 months of non-therapy amenorrhea] or surgically sterile [absence

Key Exclusion Criteria:

1. History or presence of a disease or condition that, in the Investigator's opinion, constitutes a risk when taking study drug or interfering with study assessment or interpretation of the data (e.g., autoimmune disease). Subjects post cholecystectomy are acceptable. Subjects with resolved childhood asthma not requiring prescription medicine are acceptable. Subjects with Gilbert's disease are acceptable if total bilirubin ≤3× ULN.
2. Medical history of severe allergic reaction, angioedema, anaphylaxis, clinically significant drug hypersensitivity reaction, or autoimmune or immunodeficiency disorder.
3. Active infection or a history of serious infections as follows:

   1. Use of antimicrobials (antibacterials, antivirals, antifungals, or antiparasitic agents) for an infection within 30 days before first dose. Topical treatments may be allowed at the Medical Monitor's discretion.
   2. History of opportunistic infections in the last 2 years.
   3. Recurrent or chronic infection, or other active infection, that in the opinion of the Investigator might cause this study to be detrimental to the subject.
   4. Symptomatic herpes zoster within 3 months prior to screening.
   5. History of tuberculosis (active or latent) irrespective of treatment status.
   6. Any history of viral hepatitis: hepatitis B virus, hepatitis C virus (HCV), hepatitis E virus.

      HCV is acceptable if HCV RNA is undetectable for at least 3 months post completion of direct-acting antiviral therapy.
   7. Any known history of John Cunningham virus (JCV) infection or progressive multifocal leukoencephalopathy (PML).
4. Any planned major surgical procedure during the study.
5. History of malignant neoplasm within the last 10 years, except for fully treated nonmetastatic basal or squamous cell cancers of the skin (within 3 years) that shows no evidence of recurrence.
6. Use of prescription or non-prescription drugs (including recreational drugs and herbal medications) within 7 days or 5 half-lives (whichever is longer) prior to dosing, unless in the opinion of the Investigator (in consultation with the Medical Monitor), the medication will not interfere with the study or compromise subject safety. Paracetamol (acetaminophen) at doses of ≤ 4 grams/day, and occasional use of non-steroidal anti-inflammatory drugs at licensed doses, are permitted.
7. Live or live-attenuated vaccination within 4 weeks of Day 1, or plan to receive a live vaccination during the study until follow-up.
8. Previous exposure to DR-0201, or known hypersensitivity to biologics.
9. Prior anaphylaxis to a biological agent or vaccine.
10. Neutrophil or lymphocyte counts below the normal range.
11. Estimated glomerular filtration rate by Chronic Kidney Disease Epidemiology Collaboration equation calculation ≤ 90 mL/min/1.73 m2 at screening.
12. Alanine transaminase > 2× upper limit of normal (ULN) and bilirubin > 1.5 × ULN (isolated bilirubin > 1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%) at screening. Bilirubin > 3 × ULN if known Gilbert's disease.
13. Other clinically significant abnormalities of laboratory assessments, as judged by the Investigator and/or Medical Monitor, that could affect the safety of the subject, or the interpretation of the data from the study.
14. Positive serology for human immunodeficiency virus (HIV) at screening.
15. Positive drug/alcohol screen at screening or baseline.
16. QT interval corrected for heart rate (QTc) > 450 msec, based on the mean of triplicate ECGs. The QTc is the QT interval corrected using Fridericia's formula (QTcF; preferred method), or another method, machine or overread.
17. Seated blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg at screening. Heart rate is lower than 40 bpm or higher than 100 bpm at screening.
18. Participation in a clinical trial and has received an investigational product within the following time period prior to screening in the current study: 3 months (for biologic therapies) or 1 month (for non-biologic therapies), 5 half-lives, or twice the duration of the biological effect of the investigational product (whichever is longer).
19. Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
20. Participation in a clinical study resulting in loss of blood or blood products in excess of 500 mL within 3 months prior to enrollment.
21. Any other medical or psychiatric condition, or laboratory abnormality that would, in the opinion of the Investigator or Medical Monitor, increase the subject's risk of participation, jeopardize completion of the study, or compromise interpretation of the study data. Subjects receiving systemic medication for depression are not acceptable
22. Unstable lifestyle factors (including but not limited to excessive alcohol use, heavy nicotine use, or substance abuse), to the extent that in the opinion of the Investigator they would interfere with the ability of a subject to complete the study. Up to four units of alcohol per week are allowed once the in-patient period is complete.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-11-26 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability. To determine the incidence and severity of adverse events as assessed by CTCAE v5.0 after a single IV dose | Up to 57 days

SECONDARY OUTCOMES:
PK after a single IV dose: area under the plasma concentration time curve [AUC0-t]. | Up to 57 days
PK after a single IV dose: maximum observed plasma concentration [Cmax]. | Up to 57 days
PK after a single IV dose: time of occurrence of Cmax (tmax), | Up to 57 days
PK after a single IV dose: estimated half-life | Up to 57 days

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Will, MD, Study Director — Dren Bio
Locations (1):
- Dren Investigational Site, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No